CLINICAL TRIAL: NCT02140970
Title: Double-blind, Placebo-controlled Randomized Controlled Trial of NSAID Prior to Ureteral Stent Removal in a Pediatric Population
Brief Title: Randomized Trial of NSAID vs Placebo Prior to Ureteral Stent Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-0514
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Disorder of Urinary Stent; Ureteral Spasm; Ureteropelvic Junction Obstruction; Urolithiasis
Keywords: ureteral stent; stent pain; ureteral spasm; NSAID; ibuprofen; placebo; ureteropelvic junction obstruction; urolithiasis
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral; Urolithiasis | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liquid ibuprofen (Experimental): 10 mg/kg orally up to a maximum of 400 mg given once at least 15 minutes prior to ureteral stent removal
  Interventions: Drug: Ibuprofen
- Liquid placebo (Placebo Comparator): Similar-tasting and appearing liquid placebo of equal volume to be given once orally at least 15 minutes prior to ureteral stent removal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — 10 mg/kg orally up to a maximum of 400 mg given once at least 15 minutes prior to ureteral stent removal
  Arms: Liquid ibuprofen
Drug: Placebo — Similar-tasting and appearing liquid placebo of equal volume to be given once orally at least 15 minutes prior to ureteral stent removal
  Arms: Liquid placebo

SUMMARY:
This study plans to learn more about whether ibuprofen can reduce pain after removal of a ureteral stent more than a placebo. Some patients experience pain after removal of a ureteral stent. The investigators plan to learn how often this occurs and whether it can be prevented.

The investigators hypothesize that children who have a temporary, indwelling ureteral stent will experience a significantly less post-operative pain if given a non-steroidal anti-inflammatory (NSAID) prior to removal of the ureteral stent when compared to placebo. The investigators hypothesize that the incidence of severe post-stent removal pain is similar to an adult population.

ELIGIBILITY:
Inclusion Criteria:

* ages 4-17
* unilateral ureteral stent placed after ureteropelvic junction obstruction repair or treatment of upper tract urolithiasis

Exclusion Criteria:

* bilateral stents
* undergoing other concomitant procedure at time of planned ureteral stent removal
* indication for stent other than ureteropelvic junction obstruction repair or treatment of upper tract urolithiasis
* pregnant
* developmental delay
* allergy to ibuprofen or non-steroidal anti-inflammatory medication class
* chronic kidney disease
* prior renal transplant
* history of nasal polyps
* history of asthma

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Campbell, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tadros NN, Bland L, Legg E, Olyaei A, Conlin MJ. A single dose of a non-steroidal anti-inflammatory drug (NSAID) prevents severe pain after ureteric stent removal: a prospective, randomised, double-blind, placebo-controlled trial. BJU Int. 2013 Jan;111(1):101-5. doi: 10.1111/j.1464-410X.2012.11214.x. Epub 2012 May 11. PMID 22578110

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants withdrew from the study prior to randomization.
Period: Overall Study
Arm/Group | Liquid Ibuprofen | Liquid Placebo
Started | 24 | 25
Received Intervention | 23 | 25
Analyzed | 22 | 22
Completed | 22 | 22
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Misplaced consent, subject withdrawn | 1 | 0
Not completed — Did not meet inclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only participants who were analyzed are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid Ibuprofen | Liquid Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 44
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 10.5 [4.2 to 17.3] | 12.2 [4.7 to 18.0] | 11.4 [4.2 to 18.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-operative Severe Pain (Pain Score ≥ 7)
Description: Two pain scales were used (Faces pain scale-revised [FPS-R] and visual analogue scale [VAS]) and converted to continuous value 0-10.
Time Frame: 24 hours after stent removal
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid Ibuprofen | Liquid Placebo
Number analyzed (Participants) | 22 | 22
Participants | 2 | 1

2. Secondary Outcome: Incidence of "Significantly Worsening" Pain
Description: Incidence of "significantly worsening" pain is defined as any increase ≥ 2 between the pre-operative and post-operative pain scale assessments
Time Frame: 24 hours after stent removal
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid Ibuprofen | Liquid Placebo
Number analyzed (Participants) | 22 | 22
Participants | 3 | 5

3. Secondary Outcome: Change in Pre- and Post-operative Pain Score
Description: Pain will be assessed via a 10 point [NAME OF SCALE] scale. Possible scores range from 0 to 10, with higher scores indicating more severe pain and a worse outcome.
Time Frame: 24 hours after stent removal
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Liquid Ibuprofen | Liquid Placebo
Number analyzed (Participants) | 22 | 22
score on a scale | 0.4 [-3.9 to 8] | 0.2 [-4.0 to 4.3]

4. Secondary Outcome: Opioid Usage Post-operatively
Description: This will be recorded in equivalents to milligrams intravenous morphine
Time Frame: 24 hours after stent removal
Measure: Mean (Full Range); unit: mg/kg
Arm/Group | Liquid Ibuprofen | Liquid Placebo
Number analyzed (Participants) | 22 | 22
mg/kg | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected 30 days after exposure to the intervention.
Arm/Group | Liquid Ibuprofen | Liquid Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT02140970/Prot_SAP_000.pdf